CLINICAL TRIAL: NCT01436851
Title: Nasal Provocation Testing With Nasal Lavage in Allergic and Non-allergic Occupational Rhinitis
Brief Title: Nasal Provocation Testing in Occupational Rhinitis
Acronym: NPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009/265
Record Dates: First submitted 2011-08-16; First posted 2011-09-20 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Allergic Rhinitis (Disorder)
Keywords: rhinitis; allergy; occupational; storage mites; nasal lavage; challenge test; ECP; alfa2Macroglobuline
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Participants with storage mite sensitization were challenged with placebo extract and storage mite extract in the nose.
Masking Description: The participants were challenged on two occasions, one with placebo extract, and the other with storage mite extract, but in random order, and without the participants knowing when they received allergen or placebo
Oversight: Data Monitoring Committee: No

ARMS (1):
- Storage mite and placebo nasal challenge (Experimental): Provocation in the nose with an allergen extract of a storage mite (A. Siro or L. Destructor) and with placebo allergen extract (physiologic salt water)
  Interventions: Biological: Storage mite allergen extracts

INTERVENTIONS:
Biological: Storage mite allergen extracts — Nasal provocation with increasing doses of storage mite allergen extracts
  Other Names: Acarus Siro; Lepidoglyphus Destructor

SUMMARY:
In a previous study the investigators found that many bakery workers were sensitized to storage mites, and many had rhinitis symptoms. The role of storage mites as an occupational allergen with clinical relevance has been questioned, and the investigators wanted to investigate whether a nasal provocation with a storage mite extract would trigger symptoms and objective signs of rhinitis in bakery workers and a control group.

DETAILED DESCRIPTION:
The investigations include allergy testing with skin prick testing, and measuring of specific Immunoglobulin E (IgE) in sera, answering a questionnaire, and symptom scoring before and after provocations. The participants will be investigated one day with a placebo, and another day with the allergen extract of either Acarus Siro or Lepidoglyphus Destructor. As a measurement of nasal patency we use the nasal peak inspiratory flow meter, but also clinical scoring of nasal secretion and blockage. Indices of inflammation (ECP and alfa-Macroglobulin) will be monitored in nasal lavage.

ELIGIBILITY:
Inclusion Criteria:

* bakery workers
* > 18 years
* sensitized to a storage mite (A.Siro or L. Destructor)

Exclusion Criteria:

* pregnant or breast-feeding
* infection in upper or lower airways the last month
* nasal polyposis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Measurements of indices of inflammation in nasal lavage after specific nasal provocation with storage mite allergen | Change from baseline to 10 minutes after nasal provocation
  Indices of inflammation (alfa2-macroglobulin, eosinophil cationic protein) in nasal lavage after specific nasal provocation with storage mite allergen (Acarus Siro or Lepidoglyphus Destructor) twice, the second provocation with doubled allergen concentration

SECONDARY OUTCOMES:
Rhinitis symptoms after specific nasal provocation with storage mite allergen glyphus Destructor) | Change from baseline to 10 minutes after provocation
  Rhinitis symptoms measured by symptoms score and visual analog scale, before and after specific nasal provocation with storage mite allergen (Acarus Siro, Lepidoglyphus Destructor) twice, the second time with doubled concentration of allergen
Reduction in nasal patency measured by peak nasal inspiratory flow meter after specific nasal provocation with storage mite allergen | Change from baseline to 10 minutes after provocation
  Reduction in nasal patency measured by peak nasal inspiratory flow meter before and after specific nasal provocation with storage mite allergen (Acarus Siro, Lepidoglyphus Destructor) twice, the second time with doubled concentration of allergen
Objective signs of rhinitis assessed by rhinoscopy after specific nasal provocation with storage mite allergen | Change from baseline to 10 minutes after provocation
  Objective signs of rhinitis assessed by anterior rhinoscopy, and notified as a clinical score before and after specific nasal provocation with storage mite allergen (Acarus Siro, Lepidoglyphus Destructor) twice, second time with the doubled allergen concentration

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Storaas, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Dept. of Occupational Medicine, Haukeland University Hospital, Bergen, Norway